CLINICAL TRIAL: NCT06767631
Title: Exploratory, Longitudinal Study to Define Changes in Muscle, Tendon and Neural Properties After Botuline Neurotoxin Type a (BoNT) Treatment of Spastic Equinovarus in First-ever Stroke Patients: a Pilot Study.
Brief Title: Pilot Study on Muscle, Tendon, and Neural Changes Post-Botulinum Toxin Injections in Post-stroke Spastic Equinovarus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S68672; Trial number 2024-513158-32-00 (Other: European Medicines Agency)
Record Dates: First submitted 2024-12-27; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Spasticity; Equinovarus Foot
Keywords: Botulinum Toxins; stroke; Medial Gastrocnemius Muscle; Skeletal muscle morphology; muscle composition
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- stroke patients treated with Botulinum toxine injections for spastic equinovarus (Other): This study involves a single-arm, exploratory, longitudinal design focusing on first-time stroke patients with spastic equinovarus deformity. Participants will receive Botulinum Neurotoxin Type A (BoNT-A) injections targeting medial and lateral gastrocnemius muscle as well ass soleus muscle. The intervention aims to assess changes in muscle, tendon, and neural properties before and after treatment by using instrumented spasticity assessment and threedimensional freehand ultrasound
  Interventions: Diagnostic Test: threedimensional freehand ultrasound and instrumented spasticity assessment

INTERVENTIONS:
Diagnostic Test: threedimensional freehand ultrasound and instrumented spasticity assessment — To conduct a pilot study as guidance for a future observational study to evaluate changes in muscle, tendon and neural properties after botulinum neurotoxin-A (BoNT) treatment of spastic equinovarus in first-ever stroke patients by using Three Dimensional freehand Ultrasound (3DfUS) and Instrumented Spasticity Assessment (ISA) with the aim of optimizing treatment algorithms and long-term response in this population.

SUMMARY:
Poststroke spasticity significantly impairs function, particularly through the development of pes equinovarus. Botulinum toxin A (BoNT) injections into the medial gastrocnemius (MG) are a first-line treatment. Treatment outcomes and long-term responses to interventions can vary significantly between individual patients. Additionally, there is increasing concern about potential adverse effects on muscle morphology. Further research is essential to optimize treatment strategies and improve long-term outcomes in this population. Three-dimensional freehand ultrasound (3DfUS) and instrumented spasticity assessment (ISA) are two recently developed techniques that enable the evaluation of changes in muscle, tendon, and neural properties following BoNT injections for post-stroke spastic equinovarus. These methods hold promise for providing new insights into treatment effects. Before implementing these techniques in large-scale studies, a pilot study is required for accurate sample size calculations for a prospective observational study. This study includes a protocol for a non-blinded, non-randomized open-label longitudinal pilot study. The study was approved by the European Medicines Agency ( EU CT Number 2024-513158-32) by the University Hospitals Leuven ethical committee (ID S68672). Standard deviations and effect sizes of outcome measures obtained longitudinally with 3DfUS and ISA before and after BoNT injection into MG will inform sample size calculations for future research.

DETAILED DESCRIPTION:
TRIAL RATIONALE:

To conduct a pilot study as guidance for a future observational study to evaluate changes in muscle, tendon and neural properties after botulinum neurotoxin-A (BoNT) treatment of spastic equinovarus in first-ever stroke patients by using Three Dimensional freehand Ultrasound (3DfUS) and Instrumented Spasticity Assessment (ISA) with the aim of optimizing treatment algorithms and long-term response in this population.

TRIAL DESIGN:

Non-blinded, non-randomized open label, longitudinal pilot interventional clinical trial.

In total, 4 visits will be organised:

1. V1: Baseline visit, week 0
2. V2: Injection visit, week 5-7
3. V3: Follow-up visit, week 10-12:
4. V4: End of study visit , week 18-30

4 visits are organized according to the biological functioning of BoNT. These 4 visits also correspond to the standard clinical visits as they currently proceed when a patient is treated with BoNT. At baseline visit (week 0) and injection visit (week 6) we do not expect any changes in outcome parameters since no BoNT has been injected yet. The effect of BoNT has peak effects after 4-6 weeks and a duration of action between 2 and 6 months. At follow-up visit (week 10-12) and end-of-study visit (when BoNT is clinically elaborated, week 18-30) we expect corresponding changes in outcome parameters, respectively.

At each visit, 3DfUS measurements and ISA measurements will be performed on two muscles of both legs: 1) medial gastrocnemius muscle and 2) tibialis anterior muscle. The majority of US literature in the lower limb has focused on medial gastrocnemius. Additionally, these muscles are obvious candidates because of their functional importance in locomotion. Moreover, the medial gastrocnemius is a frequently injected muscle with BoNT, whereas tibialis anterior muscle is not. From a methodological perspective, both medial gastrocnemius and tibialis anterior are superficial and can be easily tracked by means of conventional US probes and EMG electrodes.

During visit 2, a pregnancy test will be conducted prior to the injection of Botulinum toxin. If the test is positive, the study will be discontinued, and the patient will not be treated with Botulinum toxin A.

Total duration of one visit will be 1.5 to 2 hours. All measurements of one visit take place on the same day. Measurements will be performed at the University Hospital Leuven.

For this study, stroke patients treated with BoNT for spastic equinovarus will be included. In particular stroke patients are patients that are being treated at the University Hospital, Leuven. The annual number of stroke patients seen in UZ Leuven is approximately 600 per year.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
* 2. At least 18 years of age at the time of signing the Informed Consent Form (ICF)
* 3. Use of highly effective methods of birth control; defined as those that, alone or in combination, result in low failure rate (i.e., less than 1% per year) when used consistently and correctly; such as implants, injectables, combined oral contraceptives, some IUDs, true sexual abstinence (i.e. refraining from heterosexual intercourse during the entire period of risk associated with the Trial treatment(s)) or commitment to a vasectomised partner.
* 4. Pes equinovarus due to spasticity
* 5. Clinical need for BoNT injection at the lower leg
* 6. Any previous injection of BoNT into the muscles to be investigated was at least 3 months ago
* 7. First-ever, unilateral stroke

Exclusion Criteria:

* Musculoskeletal or other neurological problems affecting the lower limb
* Presence of spinal cord pathology that could lead to spasticity, ataxia, dystonia
* Cognitive problems that impede measurements
* Severe co-morbidities
* Irritated skin or open wounds where ultrasound will be placed
* Pregnancy
* Profound atrophy of the muscles in the target area(s) of injection
* Participation in an interventional Trial with an investigational medicinal product (IMP) or device
* The effect of botulinum toxin A can theoretically be potentiated by agents affecting neuromuscular transmission, such as aminoglycoside antibiotics (e.g., gentamicin, tobramycin), lithium salts, cholinesterase inhibitors and tubocurarine-like muscle relaxants ((cis)atracurium, rocuronium, suxamethonium, vecuronium). Therefore, patients on whom these medications are started during the course of the trail will be excluded.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
sample size calculation | 2 years
  To estimate the number of subjects to calculate an appropriate sample size for assessing changes in muscle, tendon and neural properties after BoNT treatment of spastic equinovarus in first-ever stroke patients by using 3DfUS and ISA in a future observational study. To calculate standard deviation and effect sizes of outcome measures obtained with 3DfUS and ISA in these patients.

SECONDARY OUTCOMES:
muscle changes | 2 years
  Secondary outcome parameters measured by 3DfUS include muscle belly length for medial gastrocnemius muscle
neural changes | 2 years
  Secondary outcome parameters measured by ISA for slow stretch measured by ISA : maximal velocity of performance (Vmax [deg/s])
functional changes | 2 years
  Medical baseline data including age, gender, body mass index, time since stroke, stroke etiology, National Institute Health Stroke Scale [15], affected side, oral medication and adverse events will be collected at each visit from the patients medical file as they are part of standard of care:
muscle changes | 2 years
  Secondary outcome parameters measured by 3DfUS include tendon length for medial gastrocnemius muscle
muscle changes | 2 years
  Secondary outcome parameters measured by 3DfUS include mid-belly cross-sectional area for medial gastrocnemius muscle
muscle changes | 2 years
  Secondary outcome parameters measured by 3DfUS include muscle belly length for tibial anterior muscle
muscle changes | 2 years
  Secondary outcome parameters measured by 3DfUS mid-belly cross-sectional area for tibial anterior muscle
muscle changes | 2 years
  Secondary outcome parameters measured by 3DfUS include mean Echo Intensity for tibial anterior muscle
muscle changes | 2 years
  Secondary outcome parameters measured by 3DfUS include mean Echo Intensity for medial gastrocnemius muscle
neural changes | 2 years
  Secondary outcome parameters measured by ISA for slow stretch measured by ISA : range of motion [deg]
neural changes | 2 years
  Secondary outcome parameters measured by ISA for slow stretch measured by ISA: stiffness [Nm/deg]
neural changes | 2 years
  Secondary outcome parameters measured by ISA for slow stretch measured by ISA work [J] (area under the power-time curve).
neural changes | 2 years
  Secondary outcome parameters measured by ISA from the fast stretch: maximal velocity of performance (Vmax [deg/s])
neural changes | 2 years
  Secondary outcome parameters measured by ISA from the fast stretch: joint angle of catch [deg]
neural changes | 2 years
  Secondary outcome parameters measured by ISA from the fast stretch: angle of EMG threshold [deg]
neural changes | 2 years
  Secondary outcome parameters measured by ISA from the fast stretch: intensity of catch (power [W]; torque times angular velocity).
functional changes | 2 years
  Modified Asworth Scale
functional changes | 2 years
  Tardieu scale
functional changes | 2 years
  Barthel Index
functional changes | 2 years
  Functional Ambulation Categories
functional changes | 2 years
  the Rivermead Mobility Index
functional changes | 2 years
  Functional Independence Measure
functional changes | 2 years
  Fugl-Meyer scale
functional changes | 2 years
  Modified Rankin Scale
functional changes | 2 years
  5 Meter Timed Walking Test
functional changes | 2 years
  Motricity Index
functional changes | 2 years
  Five-Times Sit-to-Stand Test
functional changes | 2 years
  Gait analyses

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Schillebeeckx, MD, Principal Investigator — UZ Leuven campus Pellenberg, secretariaat fysische geneeskunde en revalidatie blok 5
Locations (1):
- Uz Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanssen B, De Beukelaer N, Schless SH, Cenni F, Bar-On L, Peeters N, Molenaers G, Van Campenhout A, Van den Broeck C, Desloovere K. Reliability of Processing 3-D Freehand Ultrasound Data to Define Muscle Volume and Echo-intensity in Pediatric Lower Limb Muscles with Typical Development or with Spasticity. Ultrasound Med Biol. 2021 Sep;47(9):2702-2712. doi: 10.1016/j.ultrasmedbio.2021.04.028. Epub 2021 Jun 8. PMID 34112554